CLINICAL TRIAL: NCT01882920
Title: Cytoreductive Surgery With Hyperthermic Intra-Peritoneal Chemotherapy (HIPEC) - Goal Directed Therapy vs. Standard Fluid Therapy. Prospective Randomized Study
Brief Title: Goal Directed Therapy (GDT) in Cytoreductive Surgery (CRS) and Hyperthermic Intra Peritoneal Chemotherapy (Hipec)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, M.D., Chief of Critical Area Department, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 89/10
Record Dates: First submitted 2013-06-10; First posted 2013-06-21 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Primary Peritoneal Neoplasm; Secondary Peritoneal Neoplasm
Keywords: Cytoreductive surgery; hyperthermic intraperitoneal chemotherapy; Goal directed fluid therapy
MeSH Terms: interventions — Saline Solution; Ringer's Lactate; Ringer's Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal directed therapy intravenous restricitve fluid protocol (Experimental)
  Interventions: Drug: Goal Directed Intravenous Restrictive Fluid Therapy
- Control arm (Active Comparator)
  Interventions: Drug: Conventional Intravenous Fluid therapy

INTERVENTIONS:
Drug: Goal Directed Intravenous Restrictive Fluid Therapy — Basal infusion of crystalloids (normal saline,Ringer's lactate,Ringer's solution) at 4 ml/kg/h and boluses of colloids (HES 130/0.4 ) for values of cardiac index (CI) <2.5 l/min/m2, stroke volume index (SVI) < 35 SVI ml/m2 and stroke volume variation (SVV)> 15%. In the case of CI <2.5 l/min/m2 and SVI <35 ml/m2 with SVV < 15%, an infusion with dopamine was initiated.
  Other Names: Normal Saline; Ringer's lactate; Ringer's solution; Hydroxyethyl starch 130/0,4 (HES 130,04); Automated pulse contour
  Arms: Goal directed therapy intravenous restricitve fluid protocol
Drug: Conventional Intravenous Fluid therapy — Basal infusion of crystalloid (normal saline,Ringer's lactate,Ringer's solution)variable from 4 to 12 ml/kg/hour.
  Other Names: Normal saline; Ringer's lactate; Ringer's solution
  Arms: Control arm

SUMMARY:
The aim of the study is to assess whether in cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) the use of a protocol of intravenous fluid therapy combined with goal directed fluid therapy (GDT) is associated with a significant change in morbidity, length of hospital stay and mortality compared to a standard fluid therapy. Patients undergoing CRS and hipec are randomly divided into two treatment groups. The GDT group receive fluid intravenous therapy according to a specific treatment protocol guided by monitored hemodynamic parameters assessed using the arterial pressure signal monitoring to assess stroke volume and cardiac output via an automated pulse contour analysis (Flotrac/Vigileo®); the control group receive the standard fluid therapy (crystalloid and colloid). Fluid therapy regimen is free in the control group and targeted in the GDT group. In both groups, the investigators evaluate the incidence of major abdominal and systemic complications, the total duration of hospital stay, mortality, the total amount of fluids administered, their breakdown (crystalloid/colloid) and the total number of colloid boluses administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for Cytoreductive surgery and hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

* Patients under the age of 18, patients with hemodynamically significant aortic regurgitation and heart rhythm disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
rate of abdominal complications | 90 day postoperative complication

SECONDARY OUTCOMES:
Overall Survival | 90 day overall survival

OTHER OUTCOMES:
length of hospital stay | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ester Forastiere, M.D., Principal Investigator — Regina Elena CI
Locations (1):
- Regina Elena CI, Rome, Italy